CLINICAL TRIAL: NCT02462265
Title: A Phase II, Open-Label, Single- Center Study to Assess the Activity of Oshadi D and Oshadi R in Combination With Salvage Chemotherapy for Relapsed or Refractory Acute Myeloid Leukemia (AML) or Lymphoid Leukemia (ALL) Patients
Brief Title: Oshadi D & Oshadi R Combined With Salvage Chemotherapy for Relapsed Acute Myeloid Leukemia or Lymphoid Leukemia Patients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-AM-P2-01 Version 0.1
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Acute Myeloid Leukemia; Lymphoid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphoid | interventions — Antineoplastic Agents; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 'Oshadi D & Oshadi R; salvage therapy' (Experimental): Oshadi D (180mg/tid) & Oshadi R (180mg/tid) will be administrated orally; Salvage therapy - HAM: Hi dose cytosar (5 or 6 days) and mitoxantrone (2 or 3 days) will be administrated
  Interventions: Drug: Oshadi D & Oshadi R;; Drug: salvage therapy cytosar and mitoxantrone

INTERVENTIONS:
Drug: Oshadi D & Oshadi R; — Oshadi D (180mg/TID) & Oshadi R (180mg TID) will be administrated;
  Other Names: Anti cancer agents
Drug: salvage therapy cytosar and mitoxantrone — Salvage therapy - HAM: Hi dose cytosar (5 or 6 days) and mitoxantrone (2 or 3 days)
  Other Names: anti cancer agents

SUMMARY:
The study will be a prospective open-label single-center study in previously treated patients with Acute Myeloid Leukemia (AML) or Acute Lymphoid Leukemia (ALL). Treatment efficacy and safety of the combination of Oshadi D (DNase in Oshadi carrier) and Oshadi R (RNase in Oshadi carrier) with Salvage Chemotherapy will be evaluated. Oshadi D and Oshadi R were shown to have anti-tumor activity and good safety profile.

Patients will receive Oshadi D and Oshadi R oral treatment combined with salvage chemotherapy. Patient will be evaluated throughout the study for safety and tolerance to multiple dose regimens of Oshadi D and Oshadi R.

Efficacy will be determined by percentage of bone marrow blasts assessment at day 28 post therapy initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients is diagnosed as AML or ALL
* Relapse defined as the presence of disease after the achievement of complete remission(CR). Refractory disease is defined as progression from or no response while treated with a previous line chemotherapy regimen, or progression within 30 days of last bone marrow assessment.
* Male or female ≥ 18 years of age
* Minimal performance status (ECOG 0, ≤2)
* Patients must have a measurable disease by bone marrow blast counts of > 5 % of nucleated cells.
* Written informed consent
* Adequate hepatic function (LFTs up to X4 the normal limits), renal function calculated Creatinine clearance (CrCl) for Adverse Effects of >30)
* Ability to swallow the medications.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.

Exclusion Criteria:

* Active infectious disease uncontrolled by antibiotics.
* Partially treated induction patients (i.e. day 14 non responding patients).
* Inability to receive high dose salvage chemotherapy.
* Patient with known positive HIV serology at screening.
* Female patient who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* Evidence of ongoing cardiac dysrhythmias of NCI Common Toxicity Criteria for Adverse Effects (CTCAE ) Version 3.0 grade 2.
* Pre-existing mal absorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption.
* Mental disorders.
* Inability to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of bone marrow blasts aspirate before treatment initiation and at day 28 following treatment initiation. | 28 days
  Percentage of bone marrow blasts aspirate before treatment initiation and at day 28 following treatment initiation.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 28 days
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Gatt, MD, Principal Investigator — Hadassah Medical Center, Jrusalem, Israel